CLINICAL TRIAL: NCT00099567
Title: Metabolic Syndrome, Inflammation, and Risk of Cognitive Decline
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: Paul Beeson Faculty Scholars Program (Other); University of California, San Francisco (Other)
Other Study IDs: IA0066; 1N01AG062106 (NIH); 1R01AG021918 (NIH)
Record Dates: First submitted 2004-12-16; First posted 2004-12-17 (Estimated); Last update posted 2005-11-01 (Estimated); Status verified 2004-12

CONDITIONS: Cognitive Decline
Keywords: Metabolic Syndrome; Alzheimer's Disease; Cognitive Impairment; Inflammation
MeSH Terms: conditions — Cognitive Dysfunction; Metabolic Syndrome; Alzheimer Disease; Inflammation

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine if the metabolic syndrome is a risk factor for cognitive decline and if this association is modified by inflammation.

DETAILED DESCRIPTION:
The metabolic syndrome is a clustering of several commonly occurring disorders that include abdominal obesity, high triglycerides, low HDL cholesterol, high blood pressure, and insulin resistance. This study was conducted to determine if, as hypothesized, the presence of the metabolic syndrome is associated with more cognitive decline and greater risk of developing cognitive impairment, and whether this risk is affected by the level of inflammatory markers in the blood.

This 5-year prospective observational study was conducted from 1997 to 2002 at community clinics in two locations. A total of 2632 black and white participants, aged 70 to 79 years, were recruited from the 3075 participants in the Health, Aging and Body Composition (ABC) study conducted during the same period. Participants were screened for presence of metabolic syndrome, cognitive status, inflammatory markers, and a clinic examination was administered, when the study began and at the year 3 and 5 follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 to 79
* White or Black
* Community-dwelling in Memphis, TN or Pittsburgh, PA vicinity
* Well-functioning (no difficulty in walking a quarter of a mile or going up 10 steps without resting)

Exclusion Criteria:

* Any difficulty with activities of daily living
* Clinical dementia
* Inability to communicate with interviewer
* Intention of moving out of vicinity in the next year
* Active treatment for cancer in the previous 3 years
* Participation in a trial involving a lifestyle intervention

Ages: 70 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 2632
Dates: Start 1997-01; Study Completion 2002-12

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Yaffe, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Pittsburgh, Pennsylvania
  - Memphis, Tennessee

REFERENCES:
- [Background] Yaffe K, Lindquist K, Penninx BW, Simonsick EM, Pahor M, Kritchevsky S, Launer L, Kuller L, Rubin S, Harris T. Inflammatory markers and cognition in well-functioning African-American and white elders. Neurology. 2003 Jul 8;61(1):76-80. doi: 10.1212/01.wnl.0000073620.42047.d7. PMID 12847160
- [Background] Kalmijn S, Foley D, White L, Burchfiel CM, Curb JD, Petrovitch H, Ross GW, Havlik RJ, Launer LJ. Metabolic cardiovascular syndrome and risk of dementia in Japanese-American elderly men. The Honolulu-Asia aging study. Arterioscler Thromb Vasc Biol. 2000 Oct;20(10):2255-60. doi: 10.1161/01.atv.20.10.2255. PMID 11031212
- [Result] Yaffe K, Kanaya A, Lindquist K, Simonsick EM, Harris T, Shorr RI, Tylavsky FA, Newman AB. The metabolic syndrome, inflammation, and risk of cognitive decline. JAMA. 2004 Nov 10;292(18):2237-42. doi: 10.1001/jama.292.18.2237. PMID 15536110